CLINICAL TRIAL: NCT06127173
Title: Effect of Positive End Expiratory Pressure on Gastric Insufflation During Face Mask Induction of General Anesthesia in Children Undergoing Elective Surgery: A Prospective Randomized Controlled Study
Brief Title: Effect of PEEP on Gastric Insufflation During Face Mask Induction of General Anesthesia in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Collaborators: Fayoum University (Other)
Responsible Party: Principal Investigator, Khaled Abdelfattah Abdallah Sarhan, principal investigator, Asst. professor of anesthesia, Cairo university, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: D 343
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Anesthesia; Child
Keywords: ultrasound; gastric; residual; anesthesia; children
MeSH Terms: interventions — Positive-Pressure Respiration

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into three groups:
  * Group (ZEEP) with PEEP level 0 cmH2O.
  * Group (PEEP 3) with PEEP level 3 cmH2O.
  * Group (PEEP 5) with PEEP level 5 cmH2O.
Who Masked: Participant, Outcomes Assessor
Masking Description: An attending anesthesiologist will unfold the envelopes 10min before starting the procedure. The children and the sonographer will be blinded to patient group allocation. The attending anesthesiologist will not be blinded; however, he will not participate in the ultrasonography or data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- (group ZEEP) (Active Comparator): children will receive mask ventilation with PEEP level 0 cmH2O.
  Interventions: Other: Positive End Expiratory Pressure PEEP
- (group PEEP 3) (Experimental): children will receive mask ventilation with PEEP level 3 cmH2O.
  Interventions: Other: Positive End Expiratory Pressure PEEP
- (group PEEP 5) (Active Comparator): children will receive mask ventilation with PEEP level 3 cmH2O.
  Interventions: Other: Positive End Expiratory Pressure PEEP

INTERVENTIONS:
Other: Positive End Expiratory Pressure PEEP — children will receive different levels of PEEP during induction of anesthesia

SUMMARY:
The aim of our study is first to assess the effect of different PEEP levels on gastric volume using ultrasonography during induction of general anesthesia in children undergoing elective surgery

DETAILED DESCRIPTION:
Patients will be randomized into three groups:

* Group (ZEEP) with PEEP level 0 cmH2O.
* Group (PEEP 3) with PEEP level 3 cmH2O.
* Group (PEEP 5) with PEEP level 5 cmH2O. The principal investigator will create a computer-generated random table for randomization and allocation which will be numbered in sequence and will be sealed in envelopes. An attending anesthesiologist will unfold the envelopes 10min before starting the procedure. The parents and a sonographer will be blinded to patient group allocation. The attending anesthesiologist will not be blinded; however, the attending anesthesiologist will not participate in the ultrasonography or data analysis.

Anesthetic technique:

All children will undergo routine preoperative investigations: Complete blood count and coagulation profile. First, children will enter the recovery room for examination as regards the fulfillment of inclusion criteria to be in the study or to be excluded from the study. Second, the children will be included in the study will be premedicated using midazolam 0.5 mg/kg IM and IM atropine 0.2 mg /kg. Then a baseline antral area for each child lying supine will be measured by a single anesthesiologist using GE, LOGIC-e Ultrasound device with a 4-8 MHz transducer. The gastric antrum will be obtained in the sagittal or parasagittal plane between the left lobe of the liver and the pancreas, at the level of the aorta or inferior vena cava. The transducer will be tilted and rotated perpendicular to the long axis of the antrum, after having the longitudinal (D1) and anteroposterior (D2) diameters of the gastric antrum, the cross sectional areal, (CSA) will be calculated as follows:

CSA = D1x D2 x p/4 Gastric volume will be obtained by a formula based on a study by perlas.15 Stomach volume (mL) = (27 + 14.6 CSA (cm2)) - (1.28*age (years)). After that, the lungs will be divided into three regions: anterior, lateral and posterior, using the anterior and posterior axillary lines as boundaries. The ultrasound transducer will be placed perpendicular or parallel to the rib cage, and each region of the lung will be scanned bilaterally. The ultrasound probe will be first placed perpendicular to the rib cage to look for pulmonary atelectasis, and then the ultrasound probe will be placed parallel to the rib cage to take images at the most obvious point of pulmornary atelectasis. The scoring criteria will be Pulmonary consolidation score (zero- no consolidation; 1-minimal parietal consolidation; 2-small consolidation; 3-large consolidation). Pulmonary atelectasis will be defined as a pulmonary consolidation score ≥2 in any region.

Upon arrival to the operation room, standard monitors (5-lead electrocardiogram, pulse oximetry, noninvasive blood pressure monitoring, capnography) will be applied and continued all over the operation.

Intravenous cannula will be introduced after induction of anesthesia by inhalational induction with a facemask using sevoflurane 8% and oxygen 50% for all children. Then, all children will have 2-3mg /Kg of propofol, 1mcg/Kg of fentanyl and 0.4-0.6 mg /kg of rocronium. Face mask ventilation with pressure controlled ventilation using PIP 12cmH2O 16, a PEEP level according to randomization done before will be applied for 90s to all children and respiratory rate (RR) will be adjusted according to the rule, RR=24-age/2. Then, an appropriate sized endotracheal tube will be introduced. Anesthesia will be maintained using Isoflorane 1% MAC with the same parameters of mechanical ventilation during induction of anesthesia. Immediately after intubation, another measurement for gastric volume will be taken ultrasound guided as described before. Ringer Lactate solution will be infused according to the rule 4-2-1 till the end of surgery. Before awakening of the patient another measurement for pulmonary consolidation score will be taken. Then, they will be awakened as usual at the end of surgery and transferred to post anesthesia care unit (PACU).

ELIGIBILITY:
Inclusion Criteria:

Children aged1 to 12 years old American Society of Anesthesiologists (ASA) physical status I or II Children will be scheduled for elective surgery under general anesthesia.

Exclusion Criteria:

Parental refusal Children with increased risk of regurgitation Known respiratory diseases or uncorrected congenital heart disease

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2023-10-10 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Gastric residual volume immediately after intubation | 15 minutes
  ultrasound guided measurement of gastric residual volume immediately after intubation

SECONDARY OUTCOMES:
Lung Ultrasound Score | 15 minutes
  Each lung will be divided into 3 areas. For each area, a score of 0 to 3 has been assigned. Scores as follows, for any lung area: 0 indicates A-pattern (defined by the presence of only A-lines); 1, B-pattern (defined as the presence of 3 B-lines, well-spaced); 2, severe B-pattern (defined as the presence of crowded and coalescent B lines with or without consolidations limited to subpleural space); and 3, extended consolidation.
Qualitative gastric antrum score | 15 minutes
  * Grade 0 antrum: is defined as the absence of fluid content in both supine and RLD positions.
  * Grade 1 antrum: If fluid content is observed only in the RLD position, but not in the supine position.
  * Grade 2 antrum: If fluid is observed in both supine and RLD.

CONTACTS AND LOCATIONS:
Overall Officials: Khaled Sarhan, MD, Principal Investigator — Cairo University
Locations (1):
- Cairo university hospitals, kasralainy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided